CLINICAL TRIAL: NCT04633174
Title: Clinical Utilization of Sous Vide Cooking Devices in the Acute Rewarming of Frostbitten Extremities
Brief Title: Sous Vide Rewarming for Frostbitten Extremities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Nicholas Daniel, DO, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D21002
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Frostbite; Frostbite of Hand; Frostbite of Foot
MeSH Terms: conditions — Frostbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Sous vide device (Experimental): The intervention will be the use of a sous vide device to heat the water bath to 38oC, rather than the traditional methods of manual water exchanges or placing the frostbitten tissue under running water.
  Interventions: Device: Sous Vide Device (SVD)

INTERVENTIONS:
Device: Sous Vide Device (SVD) — A basin will be filled to the marked line with water from jugs at room temperature, for each frozen extremity. The sous vide device (SVD) will be attached to the distal edge of the basin. The SVD will be turned on and set to maintain the bath at a constant 38 degrees celsius for 30 minutes duration. The thermometers will be powered on continuously and the researcher will record temperatures simultaneously from each thermometer every 2 minutes. At the end of the 30 minute treatment, the SVD will be powered off and the extremity assessed by the researcher for warmth and pliability. If the extremity still feels cold or frozen, an additional 30 minutes in the water bath will commence, with subsequent reassessment. Rewarming will be considered complete when the affected tissue becomes red or purple, soft, and pliable.

SUMMARY:
The purpose of this study is to determine the efficacy of using sous vide devices for heating and maintaining the circulating warm water bath used in the rewarming of acute frostbite.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or up
* Age <17 with parent or guardian consent
* Ability to understand English
* Ability to provide consent to the study
* Acute frostbite of the hands or feet

Exclusion Criteria:

* Children under age 18 without parent or guardian
* Frostbite that has already thawed
* Frostbite of tissue other than hands or feet
* Inability to understand English
* Inability to provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Daniel, DO, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Limbs
Period: Overall Study
Arm/Group | Sous Vide Device
Started | 1; 2 Limbs
Completed | 1; 2 Limbs
Not Completed | 0; 0 Limbs

BASELINE CHARACTERISTICS:
Arm/Group | Sous Vide Device
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Limbs That Can be Rewarming Within 30 Minutes
Description: Assess if frostbitten extremities can be rewarmed in 30 minutes at 38 degrees celsius using the experimental device
Time Frame: 30 minutes
Measure: Number; unit: limbs
Units Other Than Participants: Limbs
Arm/Group | Sous Vide Device
Number analyzed (Participants) | 1
Number analyzed (Limbs) | 2
limbs | 2

2. Primary Outcome: Time to Rewarm in Minutes
Description: Measure the time required to rewarm frostbitten extremities until the extremity is reddish or purple in coloration, and soft and pliable
Time Frame: Up to 90 minutes
Measure: Mean (Full Range); unit: minutes
Units Other Than Participants: Limbs
Arm/Group | Sous Vide Device
Number analyzed (Participants) | 1
Number analyzed (Limbs) | 2
minutes | 25 [24 to 26]

3. Secondary Outcome: Ease of Use: Provider Review of the Investigational Device and Standard of Care
Description: Providers will report ease of use of the rewarming modalities by completing a survey. The survey consists of two questions requesting providers to indicate ease of use of 1) the device and 2) Standard of care (manual water bath) on a scale from 1-10, where 1 indicates easy and 10 indicated difficult.
Time Frame: Immediately after rewarming, up to 90 minutes
Population: One care provided completed a single survey to on the ease of use of the investigational device and standard of care. The results below are the actual response on the survey.
Measure: Number; unit: units on a scale
Units Other Than Participants: Care Providers
Groups:
- Manual Water Bath Management: Standard of care for rewarming of Frostbitten Extremities
Arm/Group | Sous Vide Device | Manual Water Bath Management
Number analyzed (Participants) | 1 | 1
Number analyzed (Care Providers) | 1 | 1
units on a scale | 1 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the extremity rewarming, up to 30 minutes.
Arm/Group | Sous Vide Device
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The recruitment period was limited to one winter season (Winter 2020-2021). During the recruitment period, only one patient was seen for frostbite.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT04633174/Prot_SAP_000.pdf